CLINICAL TRIAL: NCT04768400
Title: Quantitative Analysis Between Neuromuscular Blocking Agent and Motor Evoked Potential and Analysis of Risk Factors for the Coefficient of Variance of Motor Evoked Potential in Patients Undergoing Brain Tumor Removal Surgery: Population Approach
Brief Title: MEP and Neuromuscular Blocker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Dong Woo Han, Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3-2020-0511
Record Dates: First submitted 2021-02-17; First posted 2021-02-24 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rocuronium (Experimental): Neuromuscular blockade will be performed using rocuronium.
  Interventions: Drug: Arm I (MEP)

INTERVENTIONS:
Drug: Arm I (MEP) — Arm I (MEP): Motor evoked potential will be measured in various degree of the neuromuscular blockade.

SUMMARY:
It is important to predict the influence of the neuromuscular blocking agents on the motor evoked potential. Investigator will investigate the dose-response relationship between the degree of the neuromuscular blockade and the motor evoked potential in patients undergoing brain tumor surgery using the population approach. Investigator will investigate the influence of the other factors such as the impedence, reactance, muscel amount, and age on the motor evoked potential.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 years old or older, with American Society of Anesthesiologists Physical Status 1-3, and scheduled for elective brain tumor surgery under the monitoring of the motor evoked potential

Exclusion Criteria:

1. Central or peripheral neuromuscular disease
2. Sensory or motor nerve disorder
3. Allergy to propofol, remifentanil, and rocuronium
4. Patients with pacemaker

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Amplitude of the motor evoked potential | At intraoperative 0 hr from the start of the anesthetic induction
  Amplitude of the motor evoked potential will be evaluated at intraoperative 0 h from the start of the anesthetic induction.

SECONDARY OUTCOMES:
Amplitude of the motor evoked potential | At intraoperative 0 h from the opening of the dura
  Amplitude of the motor evoked potential will be evaluated at intraoperative 0 h from the opening of the dura.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea